CLINICAL TRIAL: NCT01753752
Title: Evaluation of the Corneal Residence Time of Chitosan-N-acetylcysteine Eye Drops in Patients With Dry Eye Syndrome After Single and Multiple Instillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gerhard Garhofer (Other)
Collaborators: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor-Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT291211
Record Dates: First submitted 2012-12-07; First posted 2012-12-20 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chitosan-N-acetylcystein (Experimental): Instillation into the study eye
  Interventions: Drug: Chitosan- N- Acetylcysteine eye drops
- Placebo (Placebo Comparator): Instillation into the fellow eye
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chitosan- N- Acetylcysteine eye drops
  Arms: Chitosan-N-acetylcystein
Drug: Placebo
  Arms: Placebo

SUMMARY:
In the elderly population, dry eye syndrome is a highly prevalent ocular disease. One mainstay of therapy for patients suffering from dry eye syndrome is the use of topically administered lubricants. One of the main disadvantages of the formulations currently available for the treatment of DES is the short residency time on the ocular surface, which increases the need for a frequent instillation of the lubricant.

Recently, Croma Pharma has introduced chitosan-N-acetylcysteine eye drops, designed for treatment of symptoms related to DES. Based on theoretical considerations and animal experiments, the new chitosan derivative may show an increased adhesion to mucins of the ocular surface and may therefore considerably increase the residence on the ocular surface. This, in turn, would limit the need for frequent treatment and decrease the burden for the patients.

It has been shown in recent Phase I studies that chitosan-N-acetylcysteine eye drops are safe and well tolerated after single and repeated instillation. The current study seeks to investigate the ocular residency time after a single dose and after 5 day b.i.d. treatment. For this purpose 2 cohorts are planned: In Cohort I, chitosan-N-acetylcysteine eye drops will be instilled once in one randomly chosen eye, whereas the fellow eye will receive placebo. Measurements of tear film thickness will be performed with optical coherence tomography (OCT) before instillation and 10 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 10 hours, 12 hours and 24 hours after instillation. In addition, ocular scattering of the tear film will be assessed with an Optical Quality Analysis System (OQAS) at the same timepoints. Determination of break up time (BUT) will be performed before and after instillation of the eye drops.

In Cohort II, chitosan-N-acetylcysteine eye drops will be instilled once daily in one eye and b.i.d. in the fellow eye on five consecutive days. Measurements of tear film thickness with OCT and OQAS will be performed every study day before the morning instillation and the day after the last instillation. Additionally, patients will be asked to answer the ocular surface disease index (OSDI©) on day 1 and day 6. BUT will be determined before and after instillation of the eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* History of dry eye syndrome for at least 3 months
* At least two of the following three criteria must apply: - Tear Break Up Time (BUT) < 10 seconds and/or - Schirmer I test < 7 mm and/or - at least 2 symptoms of dry eye syndrome (foreign body sensation, burning, photophobia, blurred vision, pain, itching)
* Normal ophthalmic findings except dry eye syndrome, ametropia < 6 Dpt.
* No administration of topical lubricants 24 hours before the screening examination

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the screening visit
* Symptoms of a clinically relevant illness other than dry eye in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Intake of parasympathomimetic or anti-psychotic drugs
* Diagnosis of severe dry eye by Schirmer I test < 2mm
* Difference in BUT between the two eyes of more than 4 seconds
* Wearing of contact lenses
* Glaucoma
* Treatment with corticosteroids in the 4 weeks preceding the study
* Topical treatment with any ophthalmic drug except topical lubricants in the 4 weeks preceding the study
* Ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Sjögren's syndrome
* Stevens-Johnson syndrome
* History of allergic conjunctivitis
* Ametropia ≥ 6 Dpt
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Tear Film thickness as measured with OCT - Cohort I | Before, 10 minutes (± 3 minutes), 1 hour (± 10 minutes), 2 hours (± 10minutes), 4 hours (± 10 minutes), 8 hours (± 20 minutes) 10 hours (± 20 minutes) and 12 hours (± 20 minutes) after instillation
Tear Film thickness as measured with OCT - Cohort II | change from baseline to after 6 days
  Tear film thickness will be assessed on 6 consecutive study days

SECONDARY OUTCOMES:
OSI (Objective Scattering Index) - Cohort I | Before, 10 minutes (± 3 minutes), 1 hour (± 10 minutes), 2 hours (± 10minutes), 4 hours (± 10 minutes), 8 hours (± 20 minutes) 10 hours (± 20 minutes) and 12 hours (± 20 minutes) after instillation
OSI (Objective Scattering Index) - Cohort II | change from baseline to after 6 days
  OSI will be assessed on 6 consecutive study days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria